CLINICAL TRIAL: NCT03019718
Title: Implementation of the Online Aftercare Intervention 'GSA-Online Plus' (Healthy and Without Stress at the Workplace)
Brief Title: Implementation of the Internet-based Aftercare Program 'GSA-Online Plus'
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johannes Gutenberg University Mainz (Other)
Collaborators: Deutsche Rentenversicherung (Other); Koblenz University of Applied Science (Other)
Responsible Party: Principal Investigator, Dr. Rüdiger Zwerenz, Principle Investigator, Johannes Gutenberg University Mainz
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RK-93604
Record Dates: First submitted 2017-01-06; First posted 2017-01-13 (Estimated); Last update posted 2018-03-05 (Actual); Status verified 2018-03

CONDITIONS: Implementation
Keywords: Inpatient rehabilitation; Internet-based intervention; Aftercare; Return to work; Psychodynamic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- GSA-Online plus (Experimental): Patients receive access to the internet-based aftercare program after inpatient treatment.
  Interventions: Other: GSA-Online plus

INTERVENTIONS:
Other: GSA-Online plus — A 12-week online writing intervention based on the Core Conflictual Relationship Theme Method (CCRT) with feedback provided by online therapists.

SUMMARY:
The purpose of this study is to implement the internet-based aftercare program 'GSA-Online plus' in several rehabilitation clinics with patients of different indications (psychosomatic, orthopedic and cardiovascular diseases). 'GSA-Online plus' is an internet-based aftercare program for patients with work-related problems or anxieties facing return to work after longterm sickness absence and inpatient rehabilitation. The patients have access to various exploratory and motivational videos on the study website until their inpatient rehabilitation ends. Afterwards, they start a 12-week writing intervention based on a psychotherapeutic concept, the psychodynamic 'Core Conflictual Relationship Theme Method (CCRT)'. Patients write weekly online diary entries which are answered by anonymous online therapists usually within 24 hours. In a previous randomised controlled trial the efficacy of the intervention was determined, whereas the current study focuses on the implementation and realization in a naturalistic setting (effectiveness).

ELIGIBILITY:
Inclusion Criteria:

* Referral (physician) or request (patient) to take part in the internet-based aftercare program
* Current or prospective employment within 4 weeks after inpatient rehabilitation
* Private internet access
* Informed consent
* Knowledge of the German language

Exclusion Criteria:

* Severe psychiatric or somatic disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-10-31 (Actual)

PRIMARY OUTCOMES:
Recommendation rate of 'GSA-Online plus' | study inclusion (T1)
  How often will 'GSA-Online plus' be recommended as an aftercare after inpatient rehabilitation?
Number of patients participating in 'GSA-Online plus' | 12 weeks after study inclusion (T14)
  At least 66% of patients with a corresponding recommendation should use 'GSA-Online plus' at least once.

SECONDARY OUTCOMES:
Future prospects of employment measured with the "Subjective Prognosis of Work Ability Scale" (SPE) | At study inclusion (T1) and 12 weeks later (T14)
Working ability measured with the short form of the "Work Ability Index" (WAI) | At study inclusion (T1) and 12 weeks later (T14)
Depressive symptoms measured with a subscale of the "Patient Health Questionnaire" (PHQ-9) | At study inclusion (T1) and 12 weeks later (T14)
Anxiety measured with the "General Anxiety Disorder Scale" (GAD-7) | At study inclusion (T1) and 12 weeks later (T14)
Somatic symptom burden measured with the Somatic Symptom Scale-8 (SSS-8) | At study inclusion (T1) and 12 weeks later (T14)
Psychosocial stressors measured with a subscale of the "Patient Health Questionnaire" (PHQ-10) | At study inclusion (T1) and 12 weeks later (T14)
Overall health status measured with the "EQ-5D-3L" questionnaire | At study inclusion (T1) and 12 weeks later (T14)
General capability measured with the "Sheehan-Disability Scale" | At study inclusion (T1) and 12 weeks later (T14)
Loneliness measured with the "Loneliness Scale" (LS-S) | At study inclusion (T1) and 12 weeks later (T14)
Psychological stress measured with the "Perceived Stress Scale" (PSS-4) | At study inclusion (T1) and 12 weeks later (T14)
Personal resources measured with the "Oslo Support Scale" (OSS-3) | At study inclusion (T1) and 12 weeks later (T14)
Personal resources measured with the "Brief Resilient Coping Scale" (BRCS) | At study inclusion (T1) and 12 weeks later (T14)
Regular Monitoring of self-rated health status | up to 12 weeks from study inclusion (T2-T13)
  Item drawn from the "EQ-5D-3L" questionnaire
Regular Monitoring of self-rated work ability | up to 12 weeks from study inclusion (T2-T13)
  Item drawn from the "Work Ability Index" (WAI)
Evaluation of the therapeutic feedback | up to 12 weeks from study inclusion (T2-T13)
  Two self developed items ('How satisfied are you with ... / How helpful was therapeutic feedback') on a five-point Likert scale.
Evaluation of GSA-Online+ | 12 weeks after study inclusion (T14)
  Self developed items to assess overall satisfaction with, helpfulness and utilization of GSA-Online+
Willingness to pay | 12 weeks after study inclusion (T14)
  Self developed items if and how much money participants would pay for GSA-Online+

CONTACTS AND LOCATIONS:
Overall Officials: Manfred E. Beutel, Prof. Dr., Principal Investigator — University Medical Center, Department of Psychosomatic Medicine and Psychotherapy, Johannes Gutenberg University Mainz
Locations (3):
- Germany (3):
  - Karl-Aschoff-Klinik, Bad Kreuznach, Rhineland-Palatinate
  - Drei-Burgen-Klinik Bad Muenster am Stein, Bad Kreuznach, Rhineland-Palatinate
  - Mittelrheinklinik Bad Salzig, Boppard, Rhineland-Palatinate

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zwerenz R, Bohme K, Wirth A, Labitzke N, Pachtchenko S, Beutel ME. Integration of the work-related online aftercare intervention 'GSA-online plus' (healthy and without stress at the workplace) into clinical practice: study protocol for an implementation study. BMC Health Serv Res. 2018 May 2;18(1):312. doi: 10.1186/s12913-018-2995-z. PMID 29716605
- See also: Online Aftercare Homepage — http://www.online-nachsorge.de